CLINICAL TRIAL: NCT02766387
Title: Evaluation of Correlations Between the 2 Minutes, 6 Minutes and 2 Kilometers Walk Tests in Patients With Transfemoral Amputees With a Microprocessor-controlled Prosthetic Knees
Brief Title: Evaluation of Correlations Between Different Walk Tests in Patients With Transfemoral Amputees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Diagnostic
Other Study IDs: 2016-A00054-47
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Amputation; Lower Extremity

ARMS (2):
- 2 minutes walk test (Experimental): fast walk test during 2 minutes in first and the 10 meters walk test, the 6 minutes walk test and the 2 kilometers walk test
  Interventions: Other: Evaluation of the correlation between walking speed in the 6MWT and in 2MWT, and the walking speed observed in the continuous 2km walk test and in the 10 meters walk test.
- 6 minutes walk test (Experimental): comfortable walk test during 6 minutes in first and the 10 meters walk test, the 2 minutes walk test and the 2 kilometers walk test
  Interventions: Other: Evaluation of the correlation between walking speed in the 6MWT and in 2MWT, and the walking speed observed in the continuous 2km walk test and in the 10 meters walk test.

INTERVENTIONS:
Other: Evaluation of the correlation between walking speed in the 6MWT and in 2MWT, and the walking speed observed in the continuous 2km walk test and in the 10 meters walk test.

SUMMARY:
Lower limb amputation (LLA) is a major public health problem, with significant human and financial impact. Epidemiological data remain scarce in the literature. The primary objective of the equipment of lower limb amputees is to give a walking ability and autonomy that are closest to the previous state before the amputation. About microprocessor-controlled prosthetic knees (MPKs), there are currently three in France who benefit from support by health insurance : 3C100 knee C-leg (Otto Bock HealthCare, Duderstadt, Germany), the Rheo Knee (Ossur, Reykjavik, Iceland) and knee HYBRID 1P360 (Proteor, Saint Apollinaire, France). These prostheses have the common feature of being equipped with a single-axis prosthetic knee, controlled by a microprocessor, wich allows to adapt instantly to the user's walking speed changes. They are indicated in the proximal amputations of the lower limbs from knee disarticulation included. Their prescription can only be made by a doctor of Physical Medicine and Rehabilitation. These prostheses are subject to four criteria attribution and reimbursement by the List of Products and Services Refundable (LPPR = Liste des Produits et Prestations Remboursables). This criteria are the ability to: have a walking speed greater than or equal to 4 km/h, walk 2km continuous, descend an inclined slop of 15% and to walk down the stairs step by step. These criteria must be validated after a minimum trial period of 15 days.

These attribution criteria raise the question today of how they are measured, no recommendation defining this procedure. While many standardized assessment tests of different gait parameters are available and used in clinical research, the attribution criteria are not being built in reference to these tests.

The overall objective of the study is to evaluate the diagnostic value of two simple clinical tests, the 2 and 6 minutes walk tests, to assess functional performance in patients with transfemoral amputees with a microprocessor-controlled Prosthetic Knees (MPKs).

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* to be major, with a proximal lower extremity amputation (from knee disarticulation included until hemipelvectomy)
* to have a microprocessor controlled prosthetic knee among the 3C100C-leg, the RHEO Knee or HYBRID 1P360 for over a month

Exclusion Criteria:

* unstable angina or myocardial infarction dated less than one month,
* pregnancy or breastfeeding
* acute event responsible for a restriction in walking
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2016-05; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
- The percentage of variance of the speed of the continuous 2km walk test and 10 meters walk test explained by the velocity estimated respectively by the 2MWT and the 6 MWT | 3 months